CLINICAL TRIAL: NCT06197217
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial Evaluating the Efficacy and Safety of WPV01 in Patients With Mild to Moderate COVID-19
Brief Title: Phase III Clinical Study Evaluating the Efficacy and Safety of WPV01 in Patients With Mild/Moderate COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Westlake Pharmaceuticals (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WPV01-CP-23
Record Dates: First submitted 2024-01-08; First posted 2024-01-09 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Mild to Moderate COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WPV01 (Experimental)
  Interventions: Drug: WPV01
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WPV01 — Subjects in the WPV01 group will receive WPV01 600mg orally (200mg, 3 tablets per dose), 3 times daily (TID) for 15 consecutive treatments
  Arms: WPV01
Drug: Placebo — Subjects in the Placebo group will receive WPV01 Placebo orally (3 tablets per dose), 3 times daily (TID) for 15 consecutive treatments
  Arms: Placebo

SUMMARY:
The study is a multicenter, randomized, double-blind, placebo-controlled efficacy, safety Phase III clinical trial designed to evaluate the efficacy and safety of WPV01 in patients with mild/moderate COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years at the time of signing informed consent, those with a history of COVID-19 were also eligible for enrollment in this study
* Meet the diagnostic criteria for mild or moderate COVID-19 infection according to the the Diagnostic and Treatment Program for COVID-19 Infections (Trial Tenth Edition) issued by the China Health and Wellness Commission:

  1. Positive for SARS-CoV-2 nucleic acid or positive for SARS-CoV-2 antigen in a nasopharyngeal swab specimen within 72 hours prior to randomization
  2. The onset of a COVID-19-related target symptom is less than 72 hours from randomization and the presence of at least 1 of the 5 key COVID-19-related symptoms with a severity of ≥2 points on the day of randomization
* Females of childbearing potential (details are defined in Appendix 3) Subjects must have a negative pregnancy test at Screening. Subjects will be required to use effective contraception throughout the study period beginning with the signing of the informed consent form and for 30 days after completion of the study.
* Eligible to understand the procedures and methods of this clinical trial, with full informed consent and voluntary participation by the subjects.

Exclusion Criteria:

* Known allergy to any of the ingredients in the investigational therapeutic agents
* Meet the diagnostic criteria for severe or critical COVID-19 infection according to the Diagnostic and Treatment Program for COVID-19 Infections (Trial Tenth Edition) issued by the China Health and Wellness Commission at the time of randomization.
* Within 14 days prior to randomization, the subject has received SARS-CoV-2 antiviral therapy or immunotherapy including, but not limited to, antiviral medications (e.g., interferon, raltegravir, lopinavir/ritonavir, favipiravir, ribavirin, chloroquine phosphate, arbidol, nirmatrelvir/ritonavir, molnupiravir, azulfidine, simnotrelvir/ritonavir, deuremidevir, and COVID-19 therapeutics approved during subsequent studies), corticosteroids, interleukin-1 inhibitors, interleukin-6 inhibitors, and intravenous immunoglobulins
* Within 3 days or 5 drug half-lives (whichever is longer) prior to randomization, the subject has used medications to alleviate symptoms of COVID-19: including, but not limited to, antipyretic/analgesic, cough suppressant/expectorant, compounded cold and flu remedies, antihistamines, anti-bacterials and anti-fungals
* Abnormal liver function at screening: total bilirubin ≥ 1.5 x upper limit of normal (ULN) or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 x ULN
* Being on dialysis or having a combination of moderate to severe renal insufficiency
* Immunocompromised at screening (including patients with malignant tumors, organ or bone marrow transplantation, or treatment with corticosteroids or other immunosuppressive agents)
* Chronic respiratory disease, including bronchial asthma, chronic obstructive pulmonary disease, at the time of screening
* Suspected or confirmed acute systemic infections other than COVID-19 at the time of screening
* Any comorbidity requiring surgery within 14 days prior to randomization, or any comorbidity considered life-threatening by the investigator within 30 days prior to randomization
* Patients who have received (within 30 days prior to randomization or within 5 drug half-lives, whichever is longer) or are expected to receive plasma therapy with SARS-CoV-2 monoclonal antibody or recovered COVID-19 during the study period
* Patients who have received any COVID-19 vaccine within 1 month prior to randomization
* Currently using or within 4 days post dose expected to use any drug or substance which are highly dependent on clearance via CYP3A4, MDR1, OAT1, or OAT3; used within 28 days prior to randomization or expected to use during the treatment drus with strong MDR1 inducer
* Patients who have difficulty in swallowing or history of gastrointestinal disorders that significantly affect the absorption of drugs
* Pregnant, lactating women
* Participated in other interventional clinical trials or use of experimental drugs within 1 month prior to administration;
* Patients who are judged by the investigator to be unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Time from first dose to sustained clinical recovery of 11 COVID-19 symptoms within 28 days | Day 1 to Day 28

SECONDARY OUTCOMES:
Decrease in viral load from baseline on Day 5 of treatment | Day 1 to Day 28
Percentage of subjects achieving sustained clinical recovery of 11 COVID-19 symptoms at Day 5, 9, 14, 21, and 28 | Day 1 to Day 28
Time to sustained clinical remission of 11 COVID-19 symptoms within 28 days of treatment | Day 1 to Day 28
Percentage of subjects achieving sustained clinical remission of 11 COVID-19 symptoms on Day 5, 9, 14, 21, and 28 | Day 1 to Day 28
Changes in 11 COVID-19-related symptom scores from baseline to Day 5, 9, 14, 21, and 28 | Day 1 to Day 28
Time from first dose to sustained clinical recovery of 5 key COVID-19 related symptoms within 28 days | Day 1 to Day 28
Percentage of subjects achieving sustained clinical recovery of 5 key COVID-19 related symptoms at Day 5, 9, 14, 21, and 28 | Day 1 to Day 28
Time to sustained clinical remission of 5 key COVID-19 related symptoms within 28 days | Day 1 to Day 28
Changes in 5 key COVID-19-related symptom scores from baseline to Day 5, 9, 14, 21, and 28 | Day 1 to Day 28
Percentage of subjects who experienced COVID-19 progression within 28 days | Day 1 to Day 28
Proportion of subjects requiring supplemental oxygen within 28 days | Day 1 to Day 28
Change in World Health Organization (WHO) Clinical Progress Scale Score within 28 days | Day 1 to Day 28
Time from first dose to SARS-CoV-2 RNA below the threshold after treatment within 14 days | Day 1 to Day 14
Percentage of subjects with SARS-CoV-2 RNA below the threshold on Day 3, 5, 7, 9 and 14 | Day 1 to Day 14
Change from baseline in viral load at each visit from treatment to Day 14 | Day 1 to Day 14
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- China Japan Friendship Hospital, Beijing, Beijing Municipality, China